CLINICAL TRIAL: NCT03439137
Title: A Phase III, Double Blind, Confirmatory Study of MT-6548 Compared to Darbepoetin Alfa in Hemodialysis Subjects With Anemia Associated With Chronic Kidney Disease in Japan
Brief Title: Efficacy and Safety Study to Evaluate MT-6548 in Hemodialysis Subjects Currently Receiving ESAs With Anemia Associated With Chronic Kidney Disease in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-6548-J03
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Results first posted 2021-04-12 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Anemia; Hemodialysis Dependent Chronic Kidney Disease
MeSH Terms: conditions — Anemia | interventions — vadadustat; Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MT-6548 (Experimental)
  Interventions: Drug: MT-6548; Drug: Darbepoetin alfa-matching placebo
- Darbepoetin alfa (Active Comparator)
  Interventions: Drug: Darbepoetin alfa; Drug: MT-6548-matching placebo

INTERVENTIONS:
Drug: MT-6548 — Oral tablet
  Other Names: vadadustat; AKB-6548
  Arms: MT-6548
Drug: Darbepoetin alfa — Intravenous administration
  Arms: Darbepoetin alfa
Drug: MT-6548-matching placebo — Oral tablet
  Arms: Darbepoetin alfa
Drug: Darbepoetin alfa-matching placebo — Intravenous administration
  Arms: MT-6548

SUMMARY:
For hemodialysis subjects currently receiving ESAs with anemia associated with chronic kidney disease, demonstrate non-inferiority of MT-6548 compared to darbepoetin alfa using Hb value and evaluate long-term safety of MT-6548.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CKD
* Receiving hemodialysis or hemodiafiltration 3 times a week for more than 12 weeks prior to the screening period, excluding receiving home dialysis or combination of peritoneal dialysis.
* Being treated with ESAs for the recent 8 weeks prior to the screening period
* Mean of the two screening Hb levels closest in time to the baseline visit is ≥9.5 g/dL and ≤12.0 g/dL
* Fluctuation between the two Hb levels closest in time to the baseline visit during the screening period less than 1.5 g/dL
* Serum ferritin ≥ 100 ng/mL, or TSAT ≥20% during the screening period
* Folate and vitamin B12 ≥ lower limit of normal during the screening period

Exclusion Criteria:

* Anemia due to a main cause other than CKD: sickle cell disease, myelodysplastic syndrome, bone marrow fibrosis, hematologic malignancy, hemolytic anemia, thalassemia, or pure red cell aplasia
* Active bleeding or recent blood loss within 8 weeks prior to the screening period
* RBC transfusion within 8 weeks prior to the screening period
* Received testosterone enanthate or mepitiostane within 8 weeks prior to the screening period
* AST, ALT, or total bilirubin >2.5 x upper limit of normal during the screening period
* Uncontrolled hypertension (diastolic blood pressure >110 mm Hg or systolic blood pressure >180 mm Hg) at the first day of the screening period and Day 1
* Ophthalmic examinations during the screening period correspond to either of the following criteria;

  * No available fundal findings
  * Findings indicating the presence of active fundal disease
* Severe heart failure (New York Heart Association Class IV)
* Cerebrovascular disorder or acute coronary syndrome (hospitalization due to unstable angina or myocardial infarction), requiring hospitalization due to urgent percutaneous intervention for coronary or heart failure within 12 weeks prior to the screening period
* Current or history of malignancy. History of malignancy with no recurrence for the recent 5 years is not an exclusion criterion
* New onset or recurrent event of deep vein thrombosis or pulmonary embolism within 12 weeks prior to the screening period
* Current or history of hemosiderosis or hemochromatosis
* History of prior organ transplantation or scheduled organ transplant, or prior transplantation of hematopoietic stem cell or bone marrow
* Males and females of childbearing potential who are unwilling to use an acceptable method of contraception during the designated period (Males: during the study and 90 days after the last dose, females: during study and 30 days after the last dose)
* Females who are pregnant or breast feeding, or are predicted to be pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (28):
- Japan (28):
  - Research site, Aichi
  - Research site, Chiba
  - Research site, Fukui
  - Research site, Fukuoka
  - Research site, Fukushima
  - Research site, Gunma
  - Research site, Hiroshima
  - Research site, Hokkaido
  - Research site, Hyōgo
  - Research site, Ibaraki
  - Research site, Kagawa
  - Research site, Kagoshima
  - Research site, Kanagawa
  - Research site, Kumamoto
  - Research site, Kyoto
  - Research site, Miyagi
  - Research site, Nagano
  - Research site, Nagasaki
  - Research site, Okayama
  - Research site, Okinawa
  - Research site, Osaka
  - Research site, Ōita
  - Research site, Saitama
  - Research site, Shiga
  - Research site, Shizuoka
  - Research site, Tokushma
  - Research site, Tokyo
  - Research site, Yamagata

REFERENCES:
- [Result] Nangaku M, Kondo K, Ueta K, Kokado Y, Kaneko G, Matsuda H, Kawaguchi Y, Komatsu Y. Efficacy and safety of vadadustat compared with darbepoetin alfa in Japanese anemic patients on hemodialysis: a Phase 3, multicenter, randomized, double-blind study. Nephrol Dial Transplant. 2021 Aug 27;36(9):1731-1741. doi: 10.1093/ndt/gfab055. PMID 33650630
- [Derived] Nangaku M, Ueta K, Nishimura K, Sasaki K, Hashimoto T. Factors affecting responsiveness of vadadustat in patients with anemia associated with chronic kidney disease: a post-hoc subgroup analysis of Japanese phase 3 randomized studies. Clin Exp Nephrol. 2024 May;28(5):391-403. doi: 10.1007/s10157-023-02432-z. Epub 2024 Mar 26. PMID 38530490
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Groups:
- MT-6548: MT-6548: Oral tablet. The dose was adjusted to 150-600 mg/day according to the pre-specified dose adjustment algorithm.
  Darbepoetin alfa matching placebo: Intravenous administration
- Darbepoetin Alfa: Darbepoetin alfa: Intravenous administration. The dose was adjusted to 5-180 ug/week, 2 weeks or 4 weeks according to the pre-specified dose adjustment algorithm.
  MT-6548-matching placebo: Oral tablet
Period: Overall Study
Arm/Group | MT-6548 | Darbepoetin Alfa
Started | 162 | 161
Completed | 120 | 135
Not Completed | 42 | 26
Not completed — Adverse Event | 16 | 12
Not completed — Physician Decision | 0 | 5
Not completed — Withdrawal by Subject | 14 | 4
Not completed — Conducting rescue therapy | 2 | 1
Not completed — Difficult to control Hb | 10 | 2
Not completed — Initiation of a renal transplant | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MT-6548 | Darbepoetin Alfa | Total
Number analyzed (Participants) | 162 | 161 | 323
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 68 | 129
  >=65 years | 101 | 93 | 194
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 52 | 110
  Male | 104 | 109 | 213
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian (Japanese) | 162 | 161 | 323
  Asian (Other) | 0 | 0 | 0
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Hb Level of Week 20 and Week 24
Time Frame: Up to Week 24
Population: This analysis was performed in subjects who measured Hb at least one visit after baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | MT-6548 | Darbepoetin Alfa
Number analyzed (Participants) | 160 | 160
g/dL | 10.61 [10.45 to 10.76] | 10.65 [10.50 to 10.80]

2. Secondary Outcome: Mean Hb Level of Week 48 and Week 52
Time Frame: Up to Week 52
Population: This analysis was performed in subjects who measured Hb at least one visit after baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | MT-6548 | Darbepoetin Alfa
Number analyzed (Participants) | 160 | 160
g/dL | 10.42 [10.27 to 10.56] | 10.62 [10.49 to 10.76]

3. Secondary Outcome: Hb Level at Each Assessment Time Point
Time Frame: Up to Week 52
Population: This analysis was performed only in subjects who have Hb data at each visit.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | MT-6548 | Darbepoetin Alfa
Number analyzed (Participants) | 162 | 161
g/dL
  Baseline | 10.73 [10.62 to 10.85] | 10.73 [10.62 to 10.84]
  Week 2: number analyzed (Participants) | 160 | 160
  Week 2 | 10.61 [10.49 to 10.73] | 10.85 [10.73 to 10.96]
  Week 4: number analyzed (Participants) | 157 | 159
  Week 4 | 10.38 [10.24 to 10.52] | 10.88 [10.77 to 10.99]
  Week 6: number analyzed (Participants) | 155 | 159
  Week 6 | 10.24 [10.09 to 10.40] | 10.83 [10.72 to 10.94]
  Week 8: number analyzed (Participants) | 150 | 158
  Week 8 | 10.24 [10.08 to 10.40] | 10.84 [10.74 to 10.95]
  Week 10: number analyzed (Participants) | 150 | 157
  Week 10 | 10.24 [10.06 to 10.41] | 10.86 [10.75 to 10.98]
  Week 12: number analyzed (Participants) | 147 | 157
  Week 12 | 10.43 [10.25 to 10.61] | 10.90 [10.79 to 11.01]
  Week 16: number analyzed (Participants) | 144 | 156
  Week 16 | 10.57 [10.41 to 10.73] | 10.80 [10.68 to 10.92]
  Week 20: number analyzed (Participants) | 140 | 154
  Week 20 | 10.69 [10.54 to 10.84] | 10.65 [10.52 to 10.78]
  Week 24: number analyzed (Participants) | 138 | 152
  Week 24 | 10.65 [10.50 to 10.81] | 10.63 [10.50 to 10.75]
  Week 28: number analyzed (Participants) | 132 | 150
  Week 28 | 10.58 [10.42 to 10.75] | 10.66 [10.54 to 10.78]
  Week 32: number analyzed (Participants) | 131 | 146
  Week 32 | 10.60 [10.43 to 10.76] | 10.77 [10.64 to 10.89]
  Week 36: number analyzed (Participants) | 126 | 142
  Week 36 | 10.49 [10.32 to 10.66] | 10.75 [10.61 to 10.88]
  Week 40: number analyzed (Participants) | 122 | 141
  Week 40 | 10.53 [10.37 to 10.68] | 10.67 [10.56 to 10.79]
  Week 44: number analyzed (Participants) | 118 | 139
  Week 44 | 10.54 [10.38 to 10.71] | 10.64 [10.52 to 10.76]
  Week 48: number analyzed (Participants) | 118 | 133
  Week 48 | 10.50 [10.33 to 10.66] | 10.63 [10.50 to 10.75]
  Week 52: number analyzed (Participants) | 115 | 133
  Week 52 | 10.47 [10.30 to 10.63] | 10.63 [10.52 to 10.74]
  Week 52 (LOCF): number analyzed (Participants) | 161 | 161
  Week 52 (LOCF) | 10.24 [10.08 to 10.41] | 10.61 [10.49 to 10.73]

4. Secondary Outcome: Percentage of Subjects With Hb Level at Each Assessment Time Point Within the Target Range During the Treatment Period
Time Frame: Up to Week 52
Population: This analysis was performed only in subjects who have Hb data at each visit.
Measure: Number; unit: percentage of subjects
Arm/Group | MT-6548 | Darbepoetin Alfa
Number analyzed (Participants) | 162 | 161
percentage of subjects
  Baseline | 81.5 | 78.9
  Week 2: number analyzed (Participants) | 160 | 160
  Week 2 | 75.0 | 81.3
  Week 4: number analyzed (Participants) | 157 | 159
  Week 4 | 63.7 | 83.0
  Week 6: number analyzed (Participants) | 155 | 159
  Week 6 | 58.1 | 84.3
  Week 8: number analyzed (Participants) | 150 | 158
  Week 8 | 56.0 | 85.4
  Week 10: number analyzed (Participants) | 150 | 157
  Week 10 | 56.7 | 81.5
  Week 12: number analyzed (Participants) | 147 | 157
  Week 12 | 61.9 | 86.6
  Week 16: number analyzed (Participants) | 144 | 156
  Week 16 | 68.8 | 84.6
  Week 20: number analyzed (Participants) | 140 | 154
  Week 20 | 73.6 | 74.0
  Week 24: number analyzed (Participants) | 138 | 152
  Week 24 | 75.4 | 75.7
  Week 28: number analyzed (Participants) | 132 | 150
  Week 28 | 70.5 | 77.3
  Week 32: number analyzed (Participants) | 131 | 146
  Week 32 | 73.3 | 79.5
  Week 36: number analyzed (Participants) | 126 | 142
  Week 36 | 67.5 | 78.9
  Week 40: number analyzed (Participants) | 122 | 141
  Week 40 | 77.0 | 81.6
  Week 44: number analyzed (Participants) | 118 | 139
  Week 44 | 74.6 | 85.6
  Week 48: number analyzed (Participants) | 118 | 133
  Week 48 | 72.9 | 79.7
  Week 52: number analyzed (Participants) | 115 | 133
  Week 52 | 75.7 | 86.5

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | MT-6548 | Darbepoetin Alfa
All-Cause Mortality (participants affected / at risk) | 2/162 | 1/161
Serious Adverse Events (participants affected / at risk) | 41/162 | 44/161
Other Adverse Events (participants affected / at risk) | 130/162 | 131/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-6548 (N=162) | Darbepoetin Alfa (N=161)
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 3
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 1
Coronary artery perforation (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 2
Rectal ulcer (Gastrointestinal disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Hepatic cyst infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Hydrocele male infected (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Mycotic endophthalmitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Shunt infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Haemodialysis complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Shunt blood flow excessive (Injury, poisoning and procedural complications) | 1 | 0
Shunt occlusion (Injury, poisoning and procedural complications) | 4 | 3
Shunt stenosis (Injury, poisoning and procedural complications) | 4 | 4
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urethral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 3
Facial paralysis (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 1 | 0
Thrombotic cerebral infarction (Nervous system disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Renal transplant (Surgical and medical procedures) | 0 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 2
Peripheral artery aneurysm rupture (Vascular disorders) | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MT-6548 (N=162) | Darbepoetin Alfa (N=161)
Retinal haemorrhage (Eye disorders) | 16 | 10
Constipation (Gastrointestinal disorders) | 7 | 12
Diarrhoea (Gastrointestinal disorders) | 25 | 24
Nausea (Gastrointestinal disorders) | 10 | 2
Vomiting (Gastrointestinal disorders) | 10 | 17
Seasonal allergy (Immune system disorders) | 4 | 12
Conjunctivitis (Infections and infestations) | 11 | 4
Gastroenteritis (Infections and infestations) | 10 | 1
Influenza (Infections and infestations) | 8 | 12
Nasopharyngitis (Infections and infestations) | 74 | 73
Contusion (Injury, poisoning and procedural complications) | 21 | 19
Shunt stenosis (Injury, poisoning and procedural complications) | 20 | 24
Skin abrasion (Injury, poisoning and procedural complications) | 9 | 15
Wound (Injury, poisoning and procedural complications) | 10 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 4
Headache (Nervous system disorders) | 13 | 5
Eczema (Skin and subcutaneous tissue disorders) | 10 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT03439137/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/37/NCT03439137/SAP_001.pdf